CLINICAL TRIAL: NCT05588986
Title: The Effect of Antenatal Corticosteroid Administration on Umbilical Artery Doppler Velocimetry in Pregnant Women Complicated With IUGR
Brief Title: The Effect of Antenatal Corticosteroid on Umbilical Artery Doppler Velocimetry in IUGR
Status: Completed | Type: Observational
Sponsor: Merve Demir (Other)
Collaborators: Marmara University (Other)
Responsible Party: Sponsor-Investigator, Merve Demir, Research assistant, Kocaeli University
Organization: Kocaeli University (Other)
Other Study IDs: Antenatal-IUGR
Record Dates: First submitted 2022-10-16; First posted 2022-10-20 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with IUGR: Pregnant women who received antenatal corticosteroid therapy and complicated with intrauterine growth retardation
  Interventions: Other: ultrasonography
- without IUGR: Pregnant women who received antenatal corticosteroid therapy and were not complicated by intrauterine growth retardation
  Interventions: Other: ultrasonography

INTERVENTIONS:
Other: ultrasonography — Umbilical artery Doppler evaluation by ultrasonography just before the first dose of antenatal corticosteroid, 24 hours and 48 hours after the last dose.

SUMMARY:
The purpose of this study is to evaluate the effect of antenatal corticosteroid administration on umbilical artery Doppler velocimetry measurements in pregnancies complicated by IUGR.

DETAILED DESCRIPTION:
This study was conducted with pregnant women who were likely to have preterm birth and were treated with antenatal corticosteroids. Betamethasone was used as an antenatal corticosteroid. UA Doppler measurements (PI, S/D ratio, RI) before antenatal corticosteroid administration and 24 and 48 hours after the last dose of corticosteroid administration were evaluated in pregnant groups complicated with IUGR and uncomplicated with IUGR and compared with each other.

ELIGIBILITY:
Inclusion Criteria:

pregnant women who were likely to have preterm delivery and were treated with antenatal corticosteroids.

Exclusion Criteria:

Pregnant women who had complicated pregnancy with fetal anomaly, who had multiple pregnancies, who left their pregnancy follow-up unfinished, and those under 18 years of age were excluded from the study.

Ages: 18 Years to 49 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women treated with antenatal corticosteroid due to a possible preterm delivery were divided into two groups as complicated and uncomplicated with IUGR.
Sampling Method: Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
systolic:diastolic ratio (S/D ratio) | 2018-2019
  Peak systolic velocity/end diastolic velocity
pulsatility index (PI) | 2018-2019
  Pulsatility Index (PI) = (Peak systolic velocity - end diastolic velocity)/(time averaged maximum velocity)
Resistive Index (RI) | 2018-2019
  Resistive Index (RI) = (Peak systolic velocity - end diastolic velocity)/(peak systolic velocity)

CONTACTS AND LOCATIONS:
Locations (1):
- Merve Demir, Kocaeli, Turkey (Türkiye)